CLINICAL TRIAL: NCT01236274
Title: The Risk of Myocardial Infarction in Users of Antipsychotic Agents: a CALIBER Study
Brief Title: The Risk of Myocardial Infarction in Users of Antipsychotic Agents
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University College, London (Other)
Responsible Party: Ruth Brauer, London School of Hygiene and Tropical Medicine
Other Study IDs: 10-01
Record Dates: First submitted 2010-11-05; First posted 2010-11-08 (Estimated); Last update posted 2010-11-08 (Estimated); Status verified 2010-11

CONDITIONS: Myocardial Infarction
Keywords: Myocardial Infarction; Antipsychotic agents; Self-controlled case series method; General Practice Research Database; Myocardial Ischaemia National Audit Project; CALIBER
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Antipsychotic agents AND MI: In the self-controlled case series study, patients who experienced a myocardial infarction and received an antipsychotic agent during up to standard (UTS) follow-up in the GPRD will be included and will act as their own control.
- Myocardial Infarction: In the case-control study, all cases with a first recorded occurrence of MI during up to standard (UTS) follow-up in the GPRD will be identified
- No Myocardial Infarction: In the case-control study, a control group with subjects who never experienced a myocardial infarction will be matched to cases (5:1) by age, gender, General Practitioner and registration in the GPRD on the date of MI of the case

SUMMARY:
A number of studies have suggested an association between the use of antipsychotic agents and cardiovascular mortality. However, the relationship between cardiac events and the use of antipsychotic drugs is not clear. Patients experiencing psychoses and in need for antipsychotic agents may be at a higher risk of cardiac events regardless of any effect of antipsychotic medication. Two studies have specifically investigated the association between the use of antipsychotics and the risk of cardiac events using Myocardial Infarction (MI) as an outcome measure, reporting no association and a positive association respectively. This difference in results may be explained by the use of different measures as well as study designs in both studies and because of different limitations with regard to controlling for lifestyle and medical risk factors. This study aims to assess the relationship between the risk of MI and recent exposure to antipsychotic agents by using the self-controlled case series method with which we are able to control for fixed confounders. The results of the self-controlled case series method will be compared to the results of a case-control study using the same data to compare the estimates of both methods.

DETAILED DESCRIPTION:
This study is part of the CALIBER (Cardiovascular disease research using linked bespoke studies and electronic records) programme funded over 5 years from the NIHR and Wellcome Trust. The central theme of the CALIBER research is linkage of the Myocardial Ischaemia National Audit Project (MINAP) with primary care (GPRD) and other resources. The overarching aim of CALIBER is to better understand the aetiology and prognosis of specific coronary phenotypes across a range of causal domains, particularly where electronic records provide a contribution beyond traditional studies. CALIBER has received both Ethics approval (ref 09/H0810/16) and ECC approval (ref ECC 2-06(b)/2009 CALIBER dataset).

The use of antipsychotics is associated with a rise in cardiovascular events. Previous studies investigating the effect of antipsychotic agents on the risk of Myocardial Infarction (MI) led to conflicting results with reports of either no association or a positive association. As patient populations for whom antipsychotic agents are indicated differ considerably from healthy comparison populations, confounding by indication could be substantial. Whilst confounding can be accounted for if known and measured, residual confounding remains a potential problem. This study aims to assess the relationship between the risk of MI and recent exposure to antipsychotic agents by using the self-controlled case series method with which we are able to control for fixed confounders. The results of the self-controlled case series method will be compared to the results of a case-control study using the same data to explore the role of confounding by indication.

ELIGIBILITY:
Inclusion Criteria:

* Patients in GPRD practices that agreed to linkage with the MINAP database
* Age over 18
* Self-controlled case-series: patients who received an antipsychotic agent during up to standard (UTS) follow-up in the GPRD
* Self-controlled case-series: patients who experienced a first record of MI at least 12 months after the start of UTS follow-up period in the GPRD data record

Exclusion Criteria:

* Patients will be excluded after experiencing their first MI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is comprised of patients registered at those GPRD practices that agreed to linkage with the MINAP database, and whose practices are "up to standard" according to the GPRD criteria.
  Self-controlled Case Series:
  Patients who experienced an MI and received an antipsychotic agent during up to standard (UTS) follow-up in the GPRD, will be included and will act as their own control.
  Case- control Study:
  All cases of first recorded occurrence of an MI, identified by the recording of a Read code in the GPRD within the UTS period until December 2009 will be identified. Five controls for each case will be selected matched by age, gender, General Practitioner and registration in the GPRD on the date of MI of the case.
Sampling Method: Non-Probability Sample
Enrollment: 90000 (Estimated)
Dates: Start 2010-11; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
First occurrence of a myocardial infarction recorded in the patient's medical record | Patients in the General Practice Research database (GPRD) are followed from registration until they leave the practice, die, or 31st of December 2009, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Brauer, Principal Investigator — London School of Hygiene and Tropical Medicine; Harry Hemingway, FRCP, Study Director — University College, London
Locations (1):
- London School of Hygiene and Tropical Medicine, London, United Kingdom

REFERENCES:
- See also: Related Info — http://www.caliberresearch.org/